CLINICAL TRIAL: NCT00699452
Title: The Potential of Candesartan to Retard the Progression of Aortic Stenosis Influences of Medical Therapy to the Atheroinflammatory Process in Stenotic Aortic Valves
Brief Title: The Potential of Candesartan to Retard the Progression of Aortic Stenosis
Acronym: ROCK-AS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Markku Kupari, Division of Cardiology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROCK-AS
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic stenosis; valve; candesartan
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Candesartan 8 mg/d for two weeks, then 16 mg/d until valve replacement surgery (approximately 3 months)
  Interventions: Drug: candesartan
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: candesartan — Candesartan 8 mg/d for two weeks, then 16 mg/d until valve replacement surgery (approximately 3 months)
  Other Names: Atacand
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The present study defines a blinded, randomized, placebo-controlled, prospective study, the aim of which is to determine the influence of effective treatment with Type 1 angiotensin II (Ang II) receptor (AT-1R) antagonist, using candesartan (target dose 16 mg) on stenotic aortic valves. The investigators will specifically quantify whether candesartan attenuates the key pathogenic mechanisms of aortic valve stenosis, namely inflammation, fibrosis, elastin degradation, calcification, and neovascularization.

DETAILED DESCRIPTION:
We will include in the study 120 consecutive patients with clinically significant, symptomatic aortic stenosis referred to the Helsinki University Central Hospital for consideration of valve replacement surgery. Patients who can be put on the hospital's normal waiting list for elective angiography (i.e who do not need urgent surgery) and who give their informed consent, will be randomized into two groups to start therapy with candesartan (8 mg/d for 2 weeks, and then 16 mg/d until surgery) or placebo. On average, the overall duration of the drug intervention will be 3 months, i.e., the average time in our institution from referral to surgery. In addition, patients (n=50) undergoing aortic valve replacement surgery due to aortic regurgitation caused by dilation of the aortic root will be included. This population consists of both patients with early sclerotic, i.e., pre-stenotic, changes in their aortic valves (n=30) and of patients without any sclerotic or stenotic changes in their aortic valves (n=20). The group with sclerotic changes in their aortic valves (n=30) will be divided into two groups to receive candesartan (8 mg/d 2 wk, and then 16 mg/d until surgery) (n=15) or placebo (n=15). The removed aortic valves will be examined utilizing real-time PCR, autoradiography, fluorometry, immunohistochemistry, double immunofluorescence, confocal microscopy, and enzyme immunoassays. With these techniques, several markers of inflammation, calcification, fibrosis, and the amount of lipid accumulation and oxidation of LDL in the valves will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 120 consecutive patients with clinically significant, symptomatic aortic stenosis referred to the Helsinki University Central Hospital for consideration of valve replacement surgery.

Exclusion Criteria:

* Individuals with past myocardial infarction, more than mild mitral valve disease, or previous cardiac surgery will be excluded.
* Patients with heart failure who need urgent surgery or those with hypotension (systolic blood pressure below 110 mm Hg) will be excluded.
* Patients already taking ACE inhibitors or AT-1R antagonists will be excluded from the study population.
* Other exclusion criteria include the following:

  * Complicated diabetes
  * Primary cardiomyopathy
  * Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception or have a positive serum pregnancy test
  * History of malignancy (unless a documented disease free period exceeding 5-years is present) with the exception of basal cell or squamous cell carcinoma of the skin. Women with a history of cervical dysplasia would be permitted to enter the study provided they had 3 consecutive clear Papanicolaou (Pap) smears
  * Hypothyroidism (TSH 1.5xULN)
  * History of alcohol or drug abuse within the last 5 years (this may affect compliance)
  * Unexplained creatine kinase (CK 3xULN) (To protect patient safety)
  * Serum creatinine >176 umol/L (2.0mg/dL)
  * Participation in another investigational drug study less than 4 weeks before enrolment in the study, or according to subjects local ethics committee requirements where a larger period is stipulated (to avoid potential misinterpretation of overlapping adverse events)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The degree of inflammation in stenotic aortic valves | 3-5 months

SECONDARY OUTCOMES:
The degree of calcification, lipid accumulation, and fibrosis in stenotic aortic valves | 3-5 months

CONTACTS AND LOCATIONS:
Overall Officials: Markku Kupari, MD, PhD, Principal Investigator — Division of Cardiology, Helsinki University Central Hospital
Locations (1):
- Division of Cardiology, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Helske-Suihko S, Laine M, Lommi J, Kaartinen M, Werkkala K, Kovanen PT, Kupari M. Is blockade of the Renin-Angiotensin system able to reverse the structural and functional remodeling of the left ventricle in severe aortic stenosis? J Cardiovasc Pharmacol. 2015 Mar;65(3):233-40. doi: 10.1097/FJC.0000000000000182. PMID 25469804